CLINICAL TRIAL: NCT06660420
Title: Phase 1 Dose Escalation and Expansion Study of PRAME T Cell Receptor (TCR) Engineered NK Cells in Participants With Recurrent and/or Refractory Melanoma (PRAMETIME-Mel)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0365; NCI-2024-08948 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Phase 1; Recurrent Melanoma; Refractory Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Escalation Phase (Experimental): The dose of PRAME-TCR-NK cells you receive will depend on when you join this study. Up to 5 dose levels of the study product will be tested. The first group of participants will receive the lowest dose level of the study product. Each new group will receive a higher dose of the study product than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose and recommended dose of the study product is found.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine
- Expansion Phase (Experimental): Participants will receive PRAME-TCR-NK cells at the recommended dose.All participants will receive the same dose level of fludarabine and cyclophosphamide
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: Cyclophosphamide — Given by IV
Drug: Fludarabine — Given by IV

SUMMARY:
To find the highest tolerable dose and recommended dose of PRAME-TCR-NK cells that can be given to participants with recurrent and/or refractory melanoma. The safety and tolerability of PRAME-TCR-NK cells will also be studied.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine he safety, tolerability, optimal cell dose (OCD), maximum tolerated dose (MTD), and recommended Phase 2 dose (RP2D) of PRAME-TCR-NK cells in participants with relapsed and/or refractory melanoma.

Secondary Objectives

1. To determine preliminary antitumor activity of PRAME-TCR-NK cells in participants with relapsed and/or relapsed and/or refractory melanoma.
2. To quantify the persistence of infused allogeneic donor PRAME-TCR-MK cells in the peripheral blood of the recipient.
3. To evaluate tissue and blood-based biomarkers associated with response and resistance to PRAME-TCR-NK cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years or older.
2. Participants must be willing and able to provide informed consent.
3. Participants must have HLA A*02:01.
4. Participants must have histologically documented locally advanced, unrespectable, or metastatic melanoma that is relapsed and/or refractory to immune checkpoint inhibitor (ICI) therapy including either anti-PD-1 either with or without anti-CTLA-4 blocking antibody and/or anti-LAG-3 antibody.

   During dose escalation, participants with cutaneous, mucosal, or unknown primary melanoma will be enrolled. Participants with uveal melanoma may be eligible for future enrollment into distinct cohorts during the dose confirmation phase. Participants should have received standard-of-care (SOC) therapy per standard clinical practice guidelines. Participants must not have had exposure to more than 3 prior lines of anti-PD-1 antibody-containing therapeutic regimens administered in the metastatic setting.
5. Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy 3 months.
7. Participants who received one or more prior systemic therapy are allowed for enrollment
8. A female participant is eligible to participate if at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidelines in during the study treatment period and for 6 months post PRAME-TCR-NK cell infusion. Female participants who become pregnant or suspect pregnancy must immediately notify their doctor.

   Female participants who become pregnant will be taken off the study.
9. Male participants must agree to follow the contraceptive guidelines during the study treatment period and for 6 months post PRAME-TCR-NK cell infusion. Male participants who father a child or suspect that they have fathered a child must immediately notify their doctor.
10. WOCBP must have a negative urine pregnancy test within 72 hours before the start of lymphodepleting chemotherapy. If a WOCBP has a urine pregnancy test that cannot be confirmed as negative, a serum (beta-human chorionic gonadotropin [£]-hCG]) pregnancy test will be required.
11. Participants must have measurable disease per the Response Evaluation Criteria in Solid Tumors (RECIST).
12. Participants must have adequate organ function as defined below within 10 days before the start of lymphodepleting chemotherapy:
13. Left ventricular ejection fraction >50%.
14. Adequate respiratory reserve defined as dyspnea Grade 0 or 1 and baseline oxygen saturation >92% in room air.
15. Willing to undergo mandatory blood collection and biopsies as required by the study.
16. Participants must agree not to receive a live vaccine for at least 24 months post-infusion.
17. Willing to sign consent for long-term follow-up on protocol PA17-0483 which will be signed at the same time with the clinical trial enrollment consent form.

Exclusion Criteria:

1. Pregnant, breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 6 months post PRAME-TCR-NK cell infusion.
2. Has received systemic anticancer therapy within 2 weeks or 5 half-lives, whichever is shorter, before the start of lymphodepleting chemotherapy. For participants treated with monoclonal antibodies, at least 3 weeks must have elapsed before the start of lymphodepleting chemotherapy. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 3 weeks after the last dose of the previous investigational agent.
3. Participants must have recovered from all AEs due to previous therapies to . Grade 1 or baseline. Participants with Grade 2 neuropathy, alopecia, or other non-relevant AEs may be deemed eligible at the discretion of the principal investigator (PI)/co-PIs. If a with . Grade 2 neuropathy, alopecia, or other non-relevant AEs may be deemed eligible at the discretion of the principal investigator (PI)/co-PIs. If a participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention before the start of lymphodepleting chemotherapy.
4. Has received prior radiotherapy within 2 weeks of the start of lymphodepleting chemotherapy. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine within 6 weeks prior to PRAME-TCR-NK infusion. Examples of live vaccines include but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza and COVID-19 vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines are live attenuated vaccines and are not allowed.
6. Has a diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (in doses exceeding10 mg daily of prednisone equivalent).
7. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in situ cancers.
8. Known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate if they completed radiation therapy, are clinically stable, and without the requirement of steroid treatment for at least 2 weeks prior to study enrollment.
9. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed.
10. Need for systemic immunosuppressive therapy or other physiological replacement of corticosteroids.
11. Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
12. Active infection (e.g., COVID-19, influenza, severe acute respiratory syndrome [SARS], recent sepsis). For participants recovered from infections, lymphodepletion may start after full recovery.
13. Known human immunodeficiency virus (HIV) infection, active or chronic hepatitis B or hepatitis C virus infection.
14. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participants participation for the full duration of the study, or is not in the best interest of the participants to participate, in the opinion of the treating investigator.
15. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
16. Has had an allogeneic tissue/solid organ transplant.
17. Clinically significant cardiovascular disease within 12 months before the start of lymphodepleting chemotherapy, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebrovascular event, or cardiac arrhythmia associated with hemodynamic instability. NOTE: A medically controlled arrhythmia would be permitted.
18. Prolongation of corrected QT interval using Fridericia's formula to >480 milliseconds.
19. Participants with bleeding or thrombotic disorders or at risk for severe hemorrhage. Participants with a known history of deep vein thrombosis/pulmonary embolism who are on appropriate anti-coagulation treatment are eligible.
20. Participants with LDH > 2.5-fold ULN. The evaluation should be conducted at screening.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Isabella C Glitza Oliva, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org